CLINICAL TRIAL: NCT05921630
Title: Impact of Pre-Test Information on Patient Compliance With the Spirometry Protocol: A Randomised Controlled Clinical Trial
Brief Title: Patient Compliance With the Spirometry Protocol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Gaziantep (Other)
Responsible Party: Principal Investigator, Sibel Doğru, PROFESSOR ASSİSTANT, University of Gaziantep
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: SDOGRU-001
Record Dates: First submitted 2023-06-12; First posted 2023-06-27 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: TEST COMPLIANCE
Keywords: Patient education; respiratory function tests; spirometry; test failure; lung function
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Control group (Placebo Comparator): Control group The control group was given standard routine information by the technician before spirometry.
  Interventions: Other: Education
- Leaflet group (Experimental): Information via leaflets: The subjects were given a leaflet prepared by the researchers based on literature review . The leaflet contained written and visual information about the steps of spirometry. The patients then underwent routine spirometry.
  Interventions: Other: Education
- Video (Experimental): Video-assisted education: Using a mobile phone, patients were shown a two-minute video prepared by the researchers in accordance with the guidelines that demonstrated how spirometry is performed.
  Interventions: Other: Education
- Leaflet + Video (Experimental): Education via leaflets + video: Subjects in this group were first given a leaflet and shown the video. They later underwent routine spirometry.
  Interventions: Other: Education

INTERVENTIONS:
Other: Education — Patient education before pulmonary function test

SUMMARY:
OBJECTIVE: In this study, the effect of brochure-based and video-assisted information given before spirometry on patient compliance will be evaluated.

PATIENTS AND METHODS: This is a randomized controlled clinical trial. Before the test, subjects in the intervention groups will be shown a brochure explaining the steps of the spirometry protocol and a video prepared for the same purpose. Standard routine information will be given to the control group by the technician before spirometry.

RESULTS: 450 patients will be included in the study. It will be investigated whether there is a difference in terms of test compliance between compliance status and age, gender, smoking status, presence of lung disease, spirometry indication, having spirometry for the first time and those receiving brochure, video and brochure-video information. Multivariate analyzes will be performed among the parameters found to be significant.

ELIGIBILITY:
Inclusion Criteria:

* Patients sent to the spirometry laboratory for forced vital capacity maneuver

Exclusion Criteria:

* illiterate and had communicational, hearing and visual impairment were excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Patient spirometry test compliance | One year
  We planned to increase patients' compliance with the spirometry test.

SECONDARY OUTCOMES:
Number of spirometry test repetitions | One year
  We planned to reduce the number of spirometry tests patients.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Gaziantep, Gaziantep, Turkey (Türkiye)

REFERENCES:
- [Derived] Dogru S, Aytac S, Al-Haithamy SAA, Ovayolu O, Sezgi C, Taylan M, Uyar M. Impact of pre-test information on patient compliance with the spirometry protocol: a randomized controlled clinical trial. Eur Rev Med Pharmacol Sci. 2023 Oct;27(20):9754-9761. doi: 10.26355/eurrev_202310_34147. PMID 37916339